CLINICAL TRIAL: NCT06520813
Title: Analysis and Measurement of Nail Morphology
Status: Active, not recruiting | Type: Observational
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, ANA MARIA RAYO PEREZ, Principal Investigator, University of Seville
Other Study IDs: MEDIDORUNGUEALARAYO
Record Dates: First submitted 2024-04-02; First posted 2024-07-25 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Morphology
Keywords: Nail; Measure; Curvature; Morphology

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Nail Group

SUMMARY:
It consists of measuring the nail plate in its different areas.

DETAILED DESCRIPTION:
It consists of measuring the nail plate in its different areas. This will not modify or alter the nail plate

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients
* Patients without any treatment on the nail plate

Exclusion Criteria:

* Pregnant patients
* Patients with uncontrolled systemic diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population that attends the pathology service, without randomization
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Normal length in milimeters of the nail plate | 1 year follow-up
  Analyze the normal parameters of length of the nail plate. The measurement will be carried out with an automatic caliper that will be positioned on the nail plate.
Normal width in milimeters of the nail plate | 1 year follow-up
  Analyze the normal parameters of width of the nail plate. The measurement will be carried out with an automatic caliper that will be positioned on the nail plate.
Normal curvature in degrees of the nail plate | 1 year follow-up
  Analyze the normal parameters of curvature of the nail plate. The measurement will be carried out with an automatic caliper that will be positioned on the nail plate.

CONTACTS AND LOCATIONS:
Overall Officials: RAQUEL GARCÍA DE LA PEÑA, DOCTOR, Study Director — University of Seville
Locations (1):
- Clinica Rayo, Seville, SEVILLA, Spain

IPD SHARING:
Plan to Share IPD: Undecided